CLINICAL TRIAL: NCT03387488
Title: Video Assisted Pericardioscopic Surgery: Minimal-invasive Implantation of Epimyocardial Pacemaker Leads in Humans (VAPS - A Pilot Study)
Brief Title: Video Assisted Pericardioscopic Surgery: Minimal-invasive Implantation of Epimyocardial Pacemaker Leads in Humans
Acronym: VAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-078; CIV-16-01-014366 (Other: EUDAMED)
Record Dates: First submitted 2017-12-15; First posted 2018-01-02 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-12

CONDITIONS: Dysrhythmia, Cardiac; Heart Failure; Pacemaker Electrode Infection; Hemodialysis-Induced Symptom; Bradycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): StingrayTM, Medtronic®
  Interventions: Device: StingrayTM, Medtronic®

INTERVENTIONS:
Device: StingrayTM, Medtronic® — Video- assisted pericardioscopic surgery for implanting epimyocardial pacemaker lead model 09090, Medtronic®
  Other Names: Clinical Investigational Lead Model 09090

SUMMARY:
Particularly in CRT (Cardiac Resynchronisation Therapy), limited accessibility of the coronary sinus along with its branches and the mismatch between the region of latest left ventricular (LV) contraction and an adequate epimyocardial vein frequently lead to therapy failure and might even be responsible for the 30 % non-responders, although this aspect has not been thoroughly investigated yet. Further complications such as postoperative micro- (i.e. increased thresholds) or macro-dislodgement (i.e. loss of stimulation success) of the LV electrodes are frequent complications leading to reoperation or a change of strategy. The current transthoracic epimyocardial approach via mini-thoracotomy circumvents the aforesaid obstacles and is regarded as the first-choice alternative approach. Participation in the trial would prevent patients from this invasive, transthoracic approach and at the same time allow the same degree of freedom in lead placement. Risks and complications are in this case comparable to the open surgical approach but with a lower risk of intraoperative rib fracture, postoperative pain with consecutive pulmonary hypo-ventilation and pneumonia.

Apart from the benefit of the single individual, societies benefit will include a much higher responder rate in CRT patients and less lead-associated infections. Thoracotomy with breach of the pleural cavity and single lung ventilation - a procedure that itself bears a high risk for postoperative atelectasis, pleural effusion and infection will be avoided.

In patients on hemo-dialysis and patients who suffer from an infected pacemaker-system, extravascular lead placement should be preferred. Again, the current open, transthoracic epimyocardial approach via mini-thoracotomy is regarded as the first-choice alternative approach.

Aim of this study is the validation of the feasibility of an alternative, minimal-invasive therapy method for implanting a cardiac pacemaker.

DETAILED DESCRIPTION:
Treatment:

Video- assisted pericardioscopic surgery for implanting epimyocardial pacemaker leads

Abridged Operation Protocol:

10 mm skin incision below the xiphoid process, blunt preparation towards the pericardial sac, insertion of the endoscope-carrying trocar, opening of the pericardium with endoscopic forceps, standardised inspection of the pericardial cavity, insertion of the bipolar Stingray® electrode via the endoscope working channel into pericardial space, implantation of the electrode into designated epimyocardial site under endoscopic vision, pacing measurements sensing, impedance, pacing threshold, interventricular delay (in CRT), panoramic fluoroscopy for future controls, retraction of the endoscope/trocar, subcutaneous tunnelling and connection of the respective electrode to:

* existing, infraclavicular CRT device, suture in layers, wound dressing
* a single- or dual-chamber pacemaker device implanted epigastrically, suture in layers, wound dressing

ELIGIBILITY:
Inclusion Criteria:

This study will include patients who are planned to undergo a pacemaker therapy within their regular medical care and who are eligible for an alternative approach for lead placement (minimal-invasive pericardioscopic surgery):

I. Patients fulfilling current, sophisticated criteria for cardiac resynchronisation therapy (CRT) (e.g. patients with symptomatic heart failure independent of functional class, prolonged QRS-duration (especially left bundle branch block), severely depressed systolic left ventricular function), but have a history of failed CRT lead implantation or showed insufficient resynchronization after conventional CRT treatment, OR

II. Haemodialysis patients fulfilling the criteria for an implantation of a cardiac pacemakers due to bradycardiac dysrhythmia, OR

III. Patients suffering from acute pacemaker-lead-infection, who require system-explantation and concomitant implantation of a new system

Further inclusion criteria:

1. Patients aged 18 years or above
2. Adults who are contractually capable and mentally able to understand and follow the instructions of the study personnel.
3. Signed informed consent prior to study participation.

Exclusion Criteria:

1. Euro Score II (http://www.euroscore.org/calc.html) > 20 %
2. Patients in NYHA functional class IV
3. Previous cardiac surgery / sternotomy
4. Previous pericarditis
5. Gender-independent myocardial wall thickness less than 5 mm
6. Coexisting cardiac/vessel aneurysmata
7. Patients with myocardial infarction within the last 4 weeks
8. Pregnancy and breast-feeding
9. Patients who are accommodated at judicial or official requests
10. Patients with known anomalies of the cardiac anatomy
11. Patients for whom beclometasone dipropionate is contraindicated
12. Patients with bleeding disorders and coagulopathy
13. Patients with a life expectancy below 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Operative mortality | 30 days
  The mortality will be documented as in the usual clinical routine.

SECONDARY OUTCOMES:
Moderate or severe operative complications | 7 days
  Operative complications (e.g. cardiac tamponade, severe bleeding, infection, lead dislodgement, pacing thresholds etc.) will be documented.
  Reduction of procedure-related postoperative complications, particular pulmonic complications in comparison to thoracotomy:
  * Duration of mechanical ventilation
  * Occurrence of pulmonary ventilation disorders:
  * Atelectasis
  * Pleural effusion
  * Pneumothorax
  * Postoperative pain obtained by visual analog pain scale
Adverse events | 12 months
  Adverse events will be documented
Overall survival | 12 months
  Overall survival will be documented as in the usual clinical routine.
Improvement of ejection mechanism | 12 months
  The acute and long-term effects of left-ventricular epimyocardial lead implantation/stimulation obtained by transthoracic echocardiography 1:
  Ejection fraction in percent, pre- and postoperative
Improvement of ventricle coordination | 12 months
  The acute and long-term effects of left-ventricular epimyocardial lead implantation/stimulation obtained by transthoracic echocardiography 2:
  Inter- and intraventricular delay in miliseconds, pre- and postoperative
Risk reduction of endocarditis in dialysis/infected patients | 12 months
  As compared to the literature

CONTACTS AND LOCATIONS:
Overall Officials: Nima Hatam, Dr. med., Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No